CLINICAL TRIAL: NCT02221973
Title: Effect of a Low Fat Milk Product on Serum Lipids Profile in Chinese Primary Dyslipidemia Subjects
Brief Title: Effect of a Low Fat Milk Product on Lipids Profile in Dyslipidemia Subjects
Acronym: Lipidown
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12.03.NRC
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2014-08

CONDITIONS: Primary Dyslipidemia
MeSH Terms: interventions — Sterols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- milk with 1.2g/d sterols and 8g/d hawthorn powder (Experimental)
  Interventions: Dietary Supplement: sterols and hawthorn powder
- milk with 1.8g/d sterols and 8g/d hawthorn powder (Experimental)
  Interventions: Dietary Supplement: sterols and hawthorn powder
- milk without sterols and hawthorn powder (Active Comparator)
  Interventions: Dietary Supplement: sterols and hawthorn powder

INTERVENTIONS:
Dietary Supplement: sterols and hawthorn powder — there are two dose level of sterols (1.2g/d; 1/8g/d)

SUMMARY:
The aim of LipiDown (Hawthorn + Phytosterol) clinical trial is to test the blood lipids reduction effect of plant sterols and hawthorn in milk powder in a pilot human trial: demonstrate potential to reduce total blood cholesterol more than 10% and/or total triglycerides more than 15%, as required by State food and drug administration (SFDA) regulation.

DETAILED DESCRIPTION:
The proposed clinical trial is a pilot randomized, double-blind, placebo controlled, parallel, multicenter study with three treatment groups.

The total number of 75 subjects should be enrolled to provide for a 20% dropout rate.

Subjects will be randomized into one of the following 3 groups:

* milk without sterols and hawthorn powder
* milk with 1.2g/d sterols and 8g/d hawthorn powder
* milk with 1.8g/d sterols and 8g/d hawthorn powder

The trial population will consist of female or male volunteers aged 18 - 65 years of age with primary mild to moderate hyperlipidemia documented by a serum cholesterol of 5.18-6.21mmol/L AND serum Triglycerides (TG): 1.7-5.65mmol/L , for at least 1 time tested by central laboratory in the past 2 weeks prior to recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female 18 to 65 years old (inclusive). Fasting Serum TC: 5.18-6.21mmol/L (equals to 200-241 mg/dl) AND Serum TG: 1.7-5.65mmol/L (equals to 150- 500 mg/dl) for at least 1 time tested by central laboratory in the past 2 weeks prior to recruitment.
* Primary dyslipidemia.
* The subject demonstrates an understanding of the given information and ability to record the requested data.
* Having obtained his/her informed consent

Exclusion Criteria:

* BMI above 32 kg/m2 ( morbid obesity).
* Pregnant or lactating women or intent to get pregnant.
* Menopause women on hormonal replacement therapy.
* Familial hyperlipidemia.
* Identified food allergy to dairy product or lactose intolerance.
* Severe diseases in heart, liver, kidney or hematopoietic system before admission.
* History of angina, myocardial infarction, coronary artery bypass, heart failure or other cardiovascular instability during the last 6 months.
* History of diabetes, GI, renal, pulmonary, hepatic and biliary, hypothyroidism, mental disease no self-control capacity or no articulate.
* Subject who are currently taking drugs that interfere with lipid profiles, including but not limited to statin, nicotinic acid, bile acid sequestrant, fibric acids, policosanol tablets.
* Subject who has received any anti-hyperlipidemia medication in the past 4 weeks.
* Subject who regularly takes supplements with the function of lipid reduction in the past 3 months or will take during the study (e.g. plant sterols, omega-3 fish oil, beta-glucan, nut-rich diet, soy protein, soluble oat fiber, red yeast rice or other cholesterol reducing functional ingredients).
* In-patient hyperlipidemia subjects.
* Alcohol > 3 glasses wine, or 2 beers, or 1 shot hard alcohol/day.
* Subject who cannot be expected to comply with the study procedures.
* Subject who is currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
serum concentration of Total Cholesterol (TC), | after 7 weeks of treatment.

SECONDARY OUTCOMES:
other lipid and lipoprotein parameters in serum samples that could reveal cardiovascular disease (CVD) risk etc. | at 4 and 7 weeks of treatment
  other lipid and lipoprotein parameters in serum samples
biomarkers of lipid oxidation and inflammation | after 7 weeks of treatment
  biomarkers of lipid oxidation and inflammation associated with atherogenesis in serum samples
phytosterol metabolism parameters | after 7 weeks of treatment
  phytosterol metabolism parameters in fecal samples
predictive marker for cardiovascular disease | after 7 weeks of treatment
  assess predictive marker for cardiovascular disease by non-invasive vascular screening device
safety parameters | after 7 weeks of treatment
  safety parameters

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Anzhen Hospital, Capital University of Medical Sciences, Beijing
  - Chao Yang 2nd Hospital, Beijing
  - Chui Yang Liu Hospital, Beijing